CLINICAL TRIAL: NCT01166906
Title: Pain Blocking During Drug Administration or Blood Collection With Needles
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Wangcun Jia, PhD., Research Scientist, University of California, Irvine
Other Study IDs: 20097245
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pain, Intractable
Keywords: pain blocking
MeSH Terms: conditions — Pain, Intractable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pain blocking — pain blocking

SUMMARY:
There is a gating mechanism in the dorsal horn of the spinal cord that acts to facilitate or inhibit transmission of pain signals to the brain. The gate can be closed by mechanical stimuli such as touch and vibration.

DETAILED DESCRIPTION:
The researcher develope a device that can use to reduce pain during drug administration or blood collection with needles.

ELIGIBILITY:
Inclusion Criteria:

* Receiving an injection with a needle
* Able to score the pain on a scale of 0-10 using the universal pain assessment tool, preferably 7 years of age or older

Exclusion Criteria:

* Current pregnancy
* Inability to understand and carry out instruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample,
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pain Blocking During Drug Administration or Blood Collection With Needles | up to 12 months
  Pain Blocking During Drug Administration or Blood Collection With Needles

CONTACTS AND LOCATIONS:
Overall Officials: Wangcun Jia, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical clinic, Irvine, California, United States